CLINICAL TRIAL: NCT02275936
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Parallel, Group Study of N91115 to Evaluate Safety and Pharmacokinetics in Patients With Cystic Fibrosis Homozygous for the F508del-CFTR Mutation
Brief Title: Study of N91115 in Patients With Cystic Fibrosis Homozygous F508del-CFTR Mutation
Acronym: SNO4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nivalis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N91115-1CF-03
Record Dates: First submitted 2014-10-14; First posted 2014-10-27 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Cystic Fibrosis
Keywords: N91115; Cavosonstat
MeSH Terms: conditions — Cystic Fibrosis | interventions — cavosonstat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 - 50 mg (Experimental): Every 12 hour oral dosing of N91115 for 28 days
  Interventions: Drug: N91115
- Group 2 - 100 mg (Experimental): Every 12 hour oral dosing of N91115 for 28 days
  Interventions: Drug: N91115
- Group 3 - 200 mg (Experimental): Every 12 hour oral dosing of N91115 for 28 days
  Interventions: Drug: N91115
- Group 4 - Placebo (Placebo Comparator): Every 12 hour oral dosing of placebo comparator for 28 days
  Interventions: Drug: N91115

INTERVENTIONS:
Drug: N91115 — S Nitrosoglutathione Reductase Inhibitor
  Other Names: Cavosonstat

SUMMARY:
This Phase 1b study in F508del-CFTR homozygous CF patients is being conducted to assess the safety of N91115 as the sole cystic fibrosis transmembrane conductance regulator (CFTR) modulator at doses near the expected therapeutic exposure level in preparation for Phase 2 studies of N91115 added to the CFTR modulator combination lumacaftor/ivacaftor when launched.

DETAILED DESCRIPTION:
Study procedures, frequency and timing are provided in the attached study schema. Adverse events and concomitant medication will be monitored throughout the study from informed consent signing until end of study participation. A Data Monitoring Committee (DMC) will also review unblinded safety data on a monthly basis throughout the study. Limitations on bronchodilators for pulmonary assessments prior to study drug dosing are described below except in emergent situations.

* Short acting β-agonists and anticholinergics will be held for at least 4 hours
* Long acting β-agonists dosed twice daily will be held for at least 12 hours
* Long acting β-agonists dosed once daily and long acting anticholinergics will be held for at least 24 hours

Screening (Day -28 to Day -3):

Patients will sign the informed consent and undergo procedures to determine eligibility including pregnancy testing, demographic information, medical history, and genotype by historical confirmation or blood sample confirmation (as applicable), height and weight, 12-Lead electrocardiogram (ECG), 48-hour Holter monitoring, chemistry, hematology, full physical examination, sweat chloride, smoking and alcohol history, spirometry, sputum microbiology, urinalysis and vital signs.

Day 1 Predose (Day -2 to -1) Patients will return to the clinic to reconfirm eligibility and assess any changes in medical history and pregnancy status. An abbreviated physical examination focusing on cardiovascular, pulmonary and gastrointestinal systems plus an assessment of weight will be conducted. The following will be obtained: 12-lead ECG, abbreviated physical exam, blood for DNA (optional), blood for leukocyte messenger ribonucleic acid (mRNA), blood inflammatory biomarkers, cystic fibrosis questionnaire-revised (CFQ-R), O2 Sat, patient global impression of change (PGIC), safety labs, serum pharmacokinetics (PK), spirometry, sputum microbiology, sweat chloride (SC) (if more than 2 weeks since the screening value was obtained), and vital signs. Sites may choose to perform any of these assessments on Day -2, Day -1 or Day 1 predose except for serum PK that starts Day 1 predose and vital signs that are done Day 1 predose.

Dosing and Food Intake:

Patients will take their dose of study drug every 12 hours at approximately the same time each morning and night. There are no restrictions related to food intake.

Dosing Days 1 and 2:

On Day 1, patients will be observed for at least 4 hours following the first dose of study drug. Patients return to the clinical site on Day 2 for a predose PK sample that is 24 hours after their first dose. Patients will be observed for at least 2 hours after the second dose on Day 2.

Days 3-28:

Patients self-administer study drug at approximately the same time each morning and evening with the exception that the morning doses on clinic Days 7, 14, 21 and 28, which will be administered and witnessed in the clinic.

Day 7 (Dosing in Clinic):

On Day 7, patients will return to the clinic to monitor any changes in health status and for an abbreviated physical exam, 12-Lead ECG, O2 Sat, safety labs, PK, spirometry, study drug compliance, SC and vital signs.

Day 14 (Dosing in Clinic):

On Day 14, patients will return to the clinic to monitor any changes in health status and for an abbreviated physical exam, urine pregnancy, 12-lead ECG, blood inflammatory biomarkers, CFQ-R, O2 Sat, safety labs, PK, spirometry, study drug compliance, SC and vital signs.

Day 21 (Dosing in Clinic):

On Day 21, patients will return to the clinic to monitor any changes in health status and for an abbreviated physical exam, 12-Lead ECG, O2 Sat, safety labs, PK, spirometry, study drug compliance, SC and vital signs.

Day 28 (Dosing in Clinic):

On Day 28 patients will return to the clinic to monitor any changes in health status and for an abbreviated physical exam, 12-Lead ECG, blood for DNA (optional), blood for leukocyte mRNA, blood inflammatory biomarkers, CFQ-R, urine pregnancy, O2 Sat, PGIC, safety labs, PK, spirometry, sputum microbiology, study drug compliance, SC, weight, and vital signs.

Day 42 (Final study day 2 weeks after last dose):

On Day 42 (± 2 days) study follow-up assessments include: abbreviated physical exam, blood inflammatory biomarkers, O2 Sat, PGIC, spirometry, SC, weight, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years with confirmed diagnosis of CF, homozygous for the F508del-CFTR mutation based on historical results generated by Ambry Genetics within the past two years or if unavailable, confirmed by testing done within the past 28 days
2. Sweat chloride ≥ 60 (milliequivalents) mEq/L, by quantitative pilocarpine iontophoresis test (QPIT) at screening
3. Weight ≥ 40 kg at screening
4. Forced expiratory volume (FEV1) ≥ 40% of predicted normal for age, gender, and height (Hankinson standards) pre- or post-bronchodilator value, at screening
5. Oxygen saturation by pulse oximetry ≥ 90% breathing ambient air, at screening
6. Hematology, clinical chemistry and urinalysis results with no clinically significant abnormalities that would interfere with the study assessments at screening

Exclusion Criteria:

1. Any acute infection, including acute upper or lower respiratory infections and pulmonary exacerbations that require treatment or hospitalization within 2 weeks of Study Day 1
2. Any change in chronic therapies for CF lung disease (e.g., Ibuprofen, Pulmozyme®, hypertonic saline, Azithromycin, Tobi®, Cayston®) within 4 weeks of Study Day 1
3. Blood hemoglobin < 10 g/dL at screening
4. Serum albumin < 2.5 g/dL at screening
5. Abnormal liver function defined as ≥ 3 x upper limit of normal (ULN) in 3 or more of the following: aspartate aminotransferase (AST), alanine aminotransferase (ALT), g-glutamyl transferase (GGT), alkaline phosphatase (ALP), or total bilirubin at screening
6. History of abnormal renal function (creatinine clearance < 50 mL/min using Cockcroft-Gault equation) within a year of screening
7. History, including the screening assessment, of ventricular tachycardia or other ventricular arrhythmias
8. History, including the screening assessment, of prolonged cardiac QT interval and/or QTcF (QT with Fridericia's correction) interval (> 450 msec)
9. History of solid organ or hematological transplantation
10. History of alcohol abuse or drug abuse (including cannabis, cocaine, and opioids) in the year prior to screening
11. Use of continuous (24 hr/day) or nocturnal supplemental oxygen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety assessments based on clinical evaluations, laboratory assessments, and adverse events. | 28 Days

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters of N91115 and its glucuronide metabolite in plasma | 28 Days
  Area under the curve(AUC) assessments
Pharmacokinetic (PK) parameters of N91115 and its glucuronide metabolite in plasma | 28 Days
  Maximum plasma concentration (Cmax) determinations
Pharmacokinetic (PK) parameters of N91115 and its glucuronide metabolite in plasma | 28 Days
  Ratio of parent:glucuronide metabolite

CONTACTS AND LOCATIONS:
Overall Officials: Scott Donaldson, MD, Principal Investigator — University of North Carolina
Locations (19):
- United States (19):
  - University of Alabama @ Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Children's CO, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - The New York Presbyterian Hospital, Columbia University Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital - Case Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Donaldson SH, Solomon GM, Zeitlin PL, Flume PA, Casey A, McCoy K, Zemanick ET, Mandagere A, Troha JM, Shoemaker SA, Chmiel JF, Taylor-Cousar JL. Pharmacokinetics and safety of cavosonstat (N91115) in healthy and cystic fibrosis adults homozygous for F508DEL-CFTR. J Cyst Fibros. 2017 May;16(3):371-379. doi: 10.1016/j.jcf.2017.01.009. Epub 2017 Feb 13. PMID 28209466